CLINICAL TRIAL: NCT05921591
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of IRL201104 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of IRL201104 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revolo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVLO 111-06
Record Dates: First submitted 2023-05-23; First posted 2023-06-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — IRL201104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose A IRL201104 (Experimental): IRL201104 or placebo IV on days 1 and 7
  Interventions: Drug: IRL201104; Drug: Placebo
- Dose B IRL201104 (Experimental): IRL201104 or placebo IV on days 1 and 7
  Interventions: Drug: IRL201104; Drug: Placebo
- Dose C IRL201104 (Experimental): IRL201104 or placebo IV on days 1 and 7
  Interventions: Drug: IRL201104; Drug: Placebo

INTERVENTIONS:
Drug: IRL201104 — Lyophilised powder for reconstitution for IV dosing
Drug: Placebo — Matching placebo for IRL201104

SUMMARY:
The purpose of this clinical study is to assess the safety, tolerability and pharmacokinetics of repeat doses of IRL201104 given to healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must provide signed informed consent.
* Participants must be in good general health.
* Body mass index (BMI) 18 to ≤ 30 kg/m2.
* Contraception use by men or women .

Key Exclusion Criteria:

* Clinically significant liver, kidney disease or cardiac disease.
* Active malignancy and/or history of malignancy in the past 5 years.
* Serious local or systemic infection within 30 days prior to Screening
* Any acute illness within 30 days prior to Day 1.
* Surgery, bone fracture or major musculoskeletal injury within the 3 months.
* Abnormal screening laboratory tests.
* Positive for human immunodeficiency virus (HIV) antibody or antigen.
* Positive hepatitis C virus (HCV) antibody or positive hepatitis B surface antigen (HBsAg).
* Positive result indicating active SARS-CoV-2 infection on Day -1.
* Positive urine drug screen/alcohol breath test at Screening.
* Positive Quantiferon Tuberculosis (TB) test.
* Systolic blood pressure (BP) > 150 mmHg or < 90 mmHg or diastolic BP > 90 mmHg or < 50 mmHg. Heart rate < 40 beats per minute (bpm) or > 100 bpm.
* Prolonged QT interval corrected by Fridericia's formula (QTcF) (> 450 ms for males and > 470 ms for females), cardiac arrhythmia, or any clinically significant abnormality in the resting electrocardiogram (ECG), as judged by the Investigator.
* All prescription and over-the-counter medications (including herbal medications), except for contraceptives and hormonal replacement therapy (HRT), are prohibited within 7 days prior to the first study intervention administration and throughout the entire duration of the study.
* All vaccines within 30 days prior and throughout the entire duration of the study.
* Administration of investigational product in another study within 30 days prior to the first study intervention administration, or five half-lives, whichever is longer.
* Blood donation within 30 days prior to the first study intervention administration.
* Females who are pregnant or breastfeeding.
* Failure to satisfy Investigator of fitness to participate for any other reason.
* Cigarette smokers and users of nicotine-containing products.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 28 days
  Number of subjects experiencing TEAE and number of TEAE will be summarised by treatment

SECONDARY OUTCOMES:
PK parameters of IRL201104 concentration in plasma | 28 days
  Individual plasma levels will be listed and summarized by treatment and collection timepoint.

OTHER OUTCOMES:
Incidence of treatment-emergent anti-drug antibody (ADA) responses | 28 days
  The presence of ADAs to IRL201104 will be listed and summarized by treatment group and timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Anoshie Ratnayake, MD, MPH, Study Director — Revolo Biotherapeutics
Locations (1):
- Revolo Phase I site, Los Angeles, California, United States